CLINICAL TRIAL: NCT01462591
Title: The Effects L-citrulline Supplementation on Arterial Stiffness, Wave Reflection, and Cardiac Autonomic Responses to Cold Exposure With Isometric Exercise
Brief Title: L-citrulline Supplementation & Cold Exposure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Arturo Figueroa, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HSC2011.6686
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension
Keywords: wave reflection; augmentation Index; heart rate variability; wasted left ventricular energy
MeSH Terms: conditions — Hypertension | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-citrulline (Experimental): L-citrulline (100mg/kg of body weight per day for 2 weeks)
  Interventions: Dietary Supplement: L-citrulline
- Maltodextrin (Placebo Comparator): 6g/day of placebo (maltodextrin)
  Interventions: Dietary Supplement: L-citrulline

INTERVENTIONS:
Dietary Supplement: L-citrulline — 2 weeks of L-citrulline supplementation (100mg/kg of body weight).

SUMMARY:
Cardiovascular disease (CVD) is considered the primary cause of death in the developed world. Large scale epidemiological studies indicate that prevalence of hypertension along with adverse cardiovascular events peak during the winter months. Moreover, during the winter months outdoor activities and physical stressors such as exercise have been associated with higher cardiovascular mortality when compared to other periods of the year. Although low environmental temperatures have been implicated as the triggering factor for cardiovascular complications, the mechanisms on how cold exposure increase cardiovascular morbidity and mortality remain to be elucidated. However, new research suggests that cold exposure may induce increases in cardiac sympathetic activity, endothelial damage and increased arterial stiffness of central arteries. Cardiovascular drugs including antihypertensive pharmacological agents seem to be inefficient to provide appropriate therapeutic effects during cold exposure. Therefore, it is imperative to propose alternative non-pharmacological therapies intended to prevent the detrimental effects of low environmental temperatures on cardiovascular function. Recently, oral supplementation of the amino acid L-citrulline has been proposed as an effective therapeutic adjuvant for the treatment of hypertension. L-citrulline is known to enhance the bioavailability of L-arginine levels and increase endothelial nitric oxide (NO) production, one of the main modulators of vascular tone and blood pressure (BP). L-citrulline supplementation has been shown to increase endothelial function, reduce BP, and ameliorate endothelial oxidative damage without any adverse effects. Our group has demonstrated that L-citrulline supplementation attenuates the BP response to cold exposure (the cold pressor test, CPT). These studies suggest that L-citrulline supplementation may be a feasible therapeutic aid in order to prevent cardiovascular complications associated with cold exposure. However the potential cardioprotective effects of L-citrulline supplementation during cold exposure with exercise have yet to be evaluated. It is hypothesized that L-citrulline supplementation would reduce arterial stiffness and blood pressure (BP) responses to physiological stress (cold exposure). This study may lead to the development of an adjunct therapy for the prevention and management of cardiovascular adverse events that are particularly increased during the winter months.

DETAILED DESCRIPTION:
The specific aims of the study are:

AIM 1: To determine the acute effects of cold exposure and isometric exercise, on cardiovascular hemodynamics and autonomic regulation. The working hypothesis is that the combination of cold exposure with isometric hand grip (IHG) exercise would evoke a greater acute increase in arterial stiffness, wave reflection, arterial BP and sympathetic activity than cold exposure or IHG alone. In order to test this hypothesis, the investigators will use an environmental chamber at a temperature of 4oC to perform non-invasive measurements of arterial stiffness (carotid-femoral, femoral-ankle, and brachial-ankle pulse wave velocity [PWV]), pulse wave analysis (aortic BP and augmentation index [AIx]) using applanation tonometry of the radial artery. In addition, the investigators will use continuous beat-by-beat digital BP, power spectral analysis of heart rate variability and blood pressure variability, and spontaneous BRS to evaluate autonomic function during cold exposure.

AIM 2: To examine the effects of L-citrulline supplementation on cardiovascular hemodynamics, autonomic regulation and endothelial function. The investigators will test the working hypothesis that L-citrulline supplementation for 14 days will attenuate the cardiovascular responses to physiological stress. The investigators will perform the same procedures previously specified in AIM I.

AIM 3: To determine the acute and chronic L-citrulline supplementation on endothelial function by measuring flow-mediated vasodilation, vasoactive substances, and Endothelial Progenitor Cells (EPCs). This aim will examine the working hypothesis L-citrulline will result in greater circulating levels of vasodilatory substances including nitric oxide, prostacyclin, and EPCs whereas vasoconstrictor substances endothelin-I (ET-1) will decrease. This aim will be tested by measuring serum levels of these substances before and immediately after the session at baseline and 7 days after the intervention.

Description of the study Forty individuals (20 men and 20 women) 18-35 years of age with normal resting BP (< 140/90 mmHg) will be enrolled in this study. Subjects should not be smokers, L-citrulline users or regular exercisers (defined as more than 120 min per week) in the last 6 months. The exclusion criteria will be any contraindication to exercise and medical conditions. Subjects with diverse ethnic backgrounds will be recruited from the Tallahassee metropolitan area by advertisement and direct communication.

Study design:

After completion of initial screening, cardiovascular function of eligible subjects will be evaluated at a room temperature of 4oor 23oC in random order. After baseline measurements, subjects will be randomly assigned to Placebo (Malt dextrin) or L-citrulline group for 14 days. Cardiovascular function will be evaluated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Blood pressure lower than 140/90mmHg
* Age 18 to 35 years
* BMI 20-39 kg/m2

Exclusion Criteria:

* Blood Pressure >160/100 mmHg
* Asthma
* Glaucoma
* Herpes simplex
* Uncontrolled diabetes
* Neurological disease
* Cardiovascular disease
* Inflammatory disease
* Kidney disease
* Hormone replacement therapy (HRT)
* Amino acid/vitamin supplementation\
* Corticosteroids or non-steroidal anti-inflammatory drugs
* Any drug known to affect BP or heart rate
* Glycemic control drugs
* Lipids reducing drugs
* Participants should not consume > 12 alcoholic drink/week
* Smokers
* Regular Exercisers (>1.5 hour/week).

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 6 weeks
  By measuring brachial and central (aortic and carotid) BP at rest and during physiological stress (cold exposure and handgrip test)

SECONDARY OUTCOMES:
Autonomic control of heart rate | 6 weeks
  By measuring heart rate variability at rest and during physiological stress.

CONTACTS AND LOCATIONS:
Overall Officials: Marcos A Sanchez-Gonzalez, M.D., Principal Investigator — The Florida State University
Locations (1):
- FSU College of Human Sciences, Tallahassee, Florida, United States